CLINICAL TRIAL: NCT06960837
Title: Ultrasound Simulation Case-based Workshop Implementation and Impact Assessment
Acronym: US Sim cases
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00117455
Record Dates: First submitted 2025-04-29; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Point-of-care Ultrasound; Simulation Training; Medical Education in Emergency Ultrasound
Keywords: point-of-care ultrasound; simulation training; medical education

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Emergency (EM) Physicians (Experimental): EM physicians will participate in a standardized simulation encounter during simulation days, resident conference, or faculty development sessions.
  Interventions: Behavioral: ultrasound simulation training case-based workshop during resident sim days

INTERVENTIONS:
Behavioral: ultrasound simulation training case-based workshop during resident sim days — Using the CAE Vimedix ultrasound simulator or standardized patient, a patient stem will be read or video shown to an individual participant. The participant will have 10 minutes to discuss the scenario and scan the simulator/patient. Participants will verbalize their findings and receive additional information, including diagnostic tests or point-of-care ultrasound (POCUS) videos, as they proceed through the case. They will be scored using a standardized rubric. For Objective Structured Clinical Exam (OSCE) testing, two independent raters, both with ultrasound fellowship training, one known to the participants and one unknown to the participants, will observe and rate the participant on a simulated POCUS case using the already published OSCE tool. The rater will read a brief standardized stem, and the participant will have 10 minutes to complete the station.

SUMMARY:
This study is a prospective cohort study implementing a point-of-care ultrasound (POCUS) simulation case-based workshop in emergency (EM) physicians at different training levels as an educational and competency-based assessment tool. The investigators incorporate elements of Miller's pyramid (second and third levels of "knows how" and "shows how") and the latter part of Kern's six step model framework for curriculum development (intervention implementation and student assessment, program evaluation, and feedback). The investigators will compare pre-/post-workshop knowledge and post-OSCE (Objective Structured Clinical Exam) technical skills scores. The investigators will also collect demographic data on baseline POCUS scans completed, training level, interest in ultrasound fellowship, monthly performed clinical POCUS scans, etc. The standardized simulation cases for EM POCUS training can then be generalized for use at any program globally to improve clinical training and patient care.

ELIGIBILITY:
Inclusion Criteria:

* Emergency medicine physicians

Exclusion Criteria:

* Emergency medicine nurses
* Emergency medicine technicians
* Advanced practice providers (APPs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-06 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in knowledge exam score | Baseline to 12 months
  Assessing the impact of the POCUS (point-of-care ultrasound) simulation workshop to improve training for clinical diagnostic thought processes.

SECONDARY OUTCOMES:
Ultrasound Competency Assessment Tool (UCAT) score | 12 months
  Assessing the impact of the POCUS (point-of-care ultrasound) simulation workshop to improve training for clinical diagnostic thought processes.
Number of POCUS (point-of-care ultrasound) exams performed per participant | 12 months
  Collected via electronic health records.
Change in quality assurance score | Baseline to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca G Theophanous, MD, MHSc, Principal Investigator — Duke University
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No